CLINICAL TRIAL: NCT05277857
Title: Mycobacterial Lung Diseases in Virginia: Sequencing and Clinical Determinants of Relapse and Outcome
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Eric R. Houpt, MD, Chief of the Division of Infectious Diseases and International Health, University of Virginia
Other Study IDs: IRB200232
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Nontuberculous Mycobacterial Lung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum or respiratory samples & environmental samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mycobacterial Lung Diseases in Virginia: sequencing and clinical determinants of relapse and outcome

DETAILED DESCRIPTION:
Nontuberculous mycobacterial (NTM) lung diseases, primarily due to M. avium complex (MAC), are an increasing clinical problem nationwide and now overtake domestic TB in terms of morbidity and mortality. It is also harder to treat and results in poorer outcomes despite longer drug regimens. In this project we utilize a state-wide clinical cohort of NTM lung disease patients to understand what features of the organism (such as the species or subtype or drug resistance profile), the host (such as antibiotic drug absorption), and the environment (such as household exposure to NTM) are most important in predicting clinical outcome. The sum of this research will direct future therapies and management algorithms for this difficult disease.

First, we will perform whole genome sequencing of NTM isolates to discern relapse versus reinfection and the environmental sources of acquisition. Second, we will utilize a state-wide cohort of new and prior diagnosed NTM lung disease patients, starting initial therapy to correlate clinical outcomes with NTM species, drug susceptibility, other bacterial in vitro assays, and serum drug levels.

ELIGIBILITY:
Inclusion Criteria:

* All subjects:

  * Race/ethnicity: any
  * Subject has no history of active Tuberculosis in the last 2 years.
  * NTM culture positive from respiratory specimen (sputum or bronchial lavage fluid)
  * Subject must have an available sputum sample that was taken in the last 2 years. If a sample is not available, the subject must be willing and able to provide a sputum sample.
  * Meets the following Infectious Diseases Society of America (IDSA) criteria for NTM lung disease:

    * 2 or more sputum (or 1 bronchoscopy/biopsy) cultures positive for "Mycobacterium Avium Complex" or "Mycobacterium abscessus) within the last 2 years.
    * Nodules, cavities, and/or bronchiectasis on CT scan within the past 2 years
    * If if the above data are not available, but a patient's Infectious Disease or Pulmonary physician has documented the diagnosis of NTM lung disease in their notes, this will suffice

PK subjects:

* Newly diagnosed with NTM lung disease and beginning antibiotics for NTM within the last 3 months from enrollment.
* Prior diagnosis of NTM lung disease, and starting initial therapy within the last 3 months prior to enrollment.
* Consent to pharmacokinetic testing within one month of enrollment and at six months of therapy

Exclusion Criteria:

* List the criteria for exclusion

All subjects:

* Age < 18 years
* Subject has cystic fibrosis or other inherited disorders of airway ciliary dysfunction (eg, primary ciliary dyskinesia)
* Unable to participate in follow-up requirements by phone or clinic visit

PK subjects:

• Unable to have blood drawn for pharmacokinetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observational study of patients with Nontuberculous Mycobacterial lung disease. A subset of newly and prior diagnosed NTM lung disease patients, that have started initial therapy within the last 3 months, and prior diagnosed NTM lung disease patients who have not been on therapy for at least 5 years, will be enrolled in the pharmacokinetics study (Aim 2).
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1 | 5 years
  Relapse versus reinfection: Perform whole genome sequencing of NTM isolates from lung disease patients from across Virginia to discern relapse versus reinfection and environmental sources of acquisition.

SECONDARY OUTCOMES:
Aim 2 | 5 years
  Patient outcomes: Utilizing the cohort of new and prior diagnosed NTM lung disease patients that have started initial therapy within the last 3 months from across Virginia, compare conventional drug susceptibility (MIC) versus pharmacokinetics/pharmacodynamics (PK/PD) indices in predicting NTM species-specific clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Division of Infectious Disease, Charlottesville, Virginia, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT05277857/ICF_001.pdf